CLINICAL TRIAL: NCT02414191
Title: Effect of Audit and Feedback on Physicians' Perioperative Temperature Management and Patient Outcomes: A Three-arm Cluster Randomized Controlled Trial to Compare Benchmarked and Ranked Feedback
Brief Title: Feedback on Perioperative Temperature Management and Patient Outcomes: Three-arm Trial to Compare Feedback
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 20140117-01H
Record Dates: First submitted 2015-03-19; First posted 2015-04-10 (Estimated); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Surgical Site Infections; Hypothermia
Keywords: Feedback; Temperature management; Anesthesia
MeSH Terms: conditions — Surgical Wound Infection; Hypothermia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): Participants in this study arm will receive no form of feedback.
- Benchmarked Feedback (Other): Participants in this study arm will receive benchmarked feedback regarding their perioperative temperature management.
  Interventions: Behavioral: Benchmarked Feedback
- Ranked Feedback (Other): Participants in this study arm will receive ranked feedback regarding their perioperative temperature management.
  Interventions: Behavioral: Ranked Feedback

INTERVENTIONS:
Behavioral: Benchmarked Feedback — Participants receive data, during the 6 month intervention phase, regarding their monthly temperature management performance in the form of benchmarked feedback, which is the measure of their performance in comparison the standard set by the hospital.
  Arms: Benchmarked Feedback
Behavioral: Ranked Feedback — Participants receive data, during the 6 month intervention phase, regarding their monthly temperature management performance in the form of ranked feedback, which is the measure of their performance in comparison to their peers.
  Arms: Ranked Feedback

SUMMARY:
The investigators aim to assess the impact of benchmarked and ranked feedback on anesthesiologists' perioperative temperature management and subsequent patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Staff Anesthesiologists at The Ottawa Hospital

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2018-04-06 (Actual); Study Completion 2018-04-06 (Actual)

PRIMARY OUTCOMES:
Patient peri-operative temperature | Within the 30 minutes immediately before or the 15 minutes immediately after anesthesia end time.

SECONDARY OUTCOMES:
Intraoperative warming device usage perioperative | intraoperative
Patient post-operative surgical site infection (SSI) rate | Within 30 days of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain Boet, MD, PhD, Principal Investigator — The Ottawa Hospital
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

REFERENCES:
- [Derived] Boet S, Bryson GL, Taljaard M, Pigford AA, McIsaac DI, Brehaut J, Forster A, Mohamed K, Clavel N, Pysyk C, Grimshaw JM; Canadian Perioperative Anesthesia Clinical Trials Group. Effect of audit and feedback on physicians' intraoperative temperature management and patient outcomes: a three-arm cluster randomized-controlled trial comparing benchmarked and ranked feedback. Can J Anaesth. 2018 Nov;65(11):1196-1209. doi: 10.1007/s12630-018-1205-0. Epub 2018 Aug 29. PMID 30159716